CLINICAL TRIAL: NCT04264312
Title: Beijing Center for Disease Prevention and Control
Brief Title: Baseline Investigation of Chronic Hepatitis B Viruses Infections: Who is Eligible for Treated Criteria
Status: Completed | Type: Observational
Sponsor: Wu Jiang (Other Government)
Responsible Party: Sponsor-Investigator, Wu Jiang, Director of institue for immunization and prevention of Beijing CDC, Centers for Disease Control and Prevention, China
Organization: Centers for Disease Control and Prevention, China (Other Government)
Other Study IDs: BJCDCWJ202001
Record Dates: First submitted 2020-02-04; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis B
Keywords: HBV; Antiviral Treatment Rate; China; Baseline Investigation
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through two-stage stratified cluster sampling, investigators studied the antiviral treatment rate and the main factors affecting the antiviral treatment in community chronic HBV infection-related liver disease population.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection is a major public health problem worldwide. China has the world's largest burden of HBV infection and will be a major contributor towards the global elimination of hepatitis B disease by 2030. While, the antiviral treatment rate and the main factors affecting the antiviral treatment in community chronic HBV infections is still unknown. In response to the above situation, Sampling applied a two-stage stratified cluster sampling design in 16 Districts and 331 Townships. Investigators wanted to know the one who is eligible for treated criteria based on community in 25 and over years old in Beijing.

ELIGIBILITY:
Inclusion Criteria:

* older than 25 years old;
* Residents with medical insurance coverage lived in Beijing more than 6 months .

Exclusion Criteria:

* Persons with pacemakers;
* Pregnant women;
* Persons with ascites;
* The one whose wound was not cured at the right upper abdomen

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are Residents with medical insurance who were older than 25 years and lived in Beijing more than 6 months. The population who are with pacemakers and ascites, pregnant, and whose wound was not cured at right upper abdomen were excluded.
Sampling Method: Probability Sample
Enrollment: 76220 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
HBsAg positive rate | Baseline
  Complete HBsAg tests for more than 60,000 people over the age of 25 in Beijing
Average rate of chronic hepatitis B accepting antiviral treatment | Baseline
  The one who is eligible for HBV treated criteria based on community in 25 and over years old in Beijing.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wu, Study Director — Beijing Center for Disease Prevention and Control
Locations (11):
- China (11):
  - Xicheng District Center for Disease Prevention and Control, Beijing, Beijing Municipality
  - Huairou District Center for Disease Prevention and Control, Beijing, Beijing Municipality
  - Daxing District Center for Disease Prevention and Control, Beijing, Beijing Municipality
  - Chaoyang District Center for Disease Control and Prevention, Beijing, Beijing Municipality
  - Dongcheng District Center for Disease Control and Prevention, Beijing, Beijing Municipality
  - Fengtai District Center for Disease Control and Prevention, Beijing, Beijing Municipality
  - Changping District Center for Disease Prevention and Control, Beijing
  - FangShan District Center for Disease Prevention and Control, Beijing
  - Haidian District Center for Disease Prevention and Control, Beijing
  - Miyun District Center for Disease Prevention and Control, Beijing
  - Tongzhou District Center for Disease Prevention and Control, Beijing